CLINICAL TRIAL: NCT05566795
Title: LOGGIC/FIREFLY-2: A Phase 3, Randomized, International Multicenter Trial of DAY101 Monotherapy Versus Standard of Care Chemotherapy in Patients With Pediatric Low-Grade Glioma Harboring an Activating RAF Alteration Requiring First-Line Systemic Therapy
Brief Title: DAY101 vs. Standard of Care Chemotherapy in Pediatric Participants With Low-Grade Glioma Requiring First-Line Systemic Therapy (LOGGIC/FIREFLY-2)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Day One Biopharmaceuticals, Inc. (Industry)
Collaborators: SIOPe Brain Tumor Group LOGGIC Consortium (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DAY101-002; 2022-001363-27 (EudraCT Number)
Record Dates: First submitted 2022-09-16; First posted 2022-10-04 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-11

CONDITIONS: Low-grade Glioma; Rapidly Accelerated Fibrosarcoma (RAF) Altered Glioma; Pediatric Low-grade Glioma
Keywords: Rapidly accelerated fibrosarcoma; RAF alteration glioma; Glioneural tumor; Ojemda
MeSH Terms: conditions — Noonan Syndrome 5 | interventions — tovorafenib; Antineoplastic Agents; Carboplatin

STUDY DESIGN:
Intervention Model Description: Tovorafenib versus standard of care chemotherapy
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Tovorafenib (Experimental)
  Interventions: Drug: Tovorafenib
- Investigator's choice of Standard of care therapy (Active Comparator)
  Interventions: Drug: Chemotherapeutic Agent

INTERVENTIONS:
Drug: Tovorafenib — Oral Tablet Powder for Oral Suspension
  Other Names: DAY101, Ojemda
  Arms: Tovorafenib
Drug: Chemotherapeutic Agent — Intravenous solution for injection
  Other Names: COG-V/C; SIOPe-LGG-V/C; VBL; Carboplatin
  Arms: Investigator's choice of Standard of care therapy

SUMMARY:
This is a 2-arm, randomized, open-label, multicenter, global, Phase 3 trial to evaluate the efficacy, safety, and tolerability of tovorafenib monotherapy versus standard of care (SoC) chemotherapy in participants with pediatric low-grade glioma (LGG) harboring an activating rapidly accelerated fibrosarcoma (RAF) alteration requiring first-line systemic therapy.

DETAILED DESCRIPTION:
Approximately 400 treatment-naïve LGG participants will be randomized 1:1 to either tovorafenib (Arm 1) or an Investigator's choice of SoC chemotherapy (Arm 2).

Arm 1 (tovorafenib): Treatment cycles will repeat every 28 days in the absence of disease progression. Participants will continue tovorafenib until any of the following occurs: disease progression, unacceptable toxicity, withdrawal of consent to treatment, or end of study.

Arm 2 (Investigator's Choice of SoC Chemotherapy): Participants will receive one of 4 SoC chemotherapy options selected by the treating Investigator: Children's Oncology Group - Vincristine/Carboplatin (COG-V/C) regimen, International Society for Paediatric Oncology - Low-Grade Glioma Vincristine/Carboplatin (SIOPe-LGG-V/C) regimen, vinblastine (VBL) regimen, or monthly carboplatin. The choice of SoC chemotherapy regimen will be selected prior to participant randomization. Treatment will continue until completion of therapy or until any of the following occurs: disease progression, unacceptable toxicity, withdrawal of consent to treatment, or end of study.

Participants who discontinue treatment due to disease progression will have (1) radiographic evidence of disease progression, as determined by the Investigator, or (2) clinical progression, as determined by the Investigator. Investigators are encouraged to discuss cases of clinical progression and early radiographic progression without clinical symptoms with the Sponsor Medical Monitor prior to treatment discontinuation or initiation of a different form of treatment for the malignancy. Participants may continue therapy beyond progressive disease (PD).

ELIGIBILITY:
Inclusion Criteria:

* Less than 25 years of age with LGG with known activating RAF alteration.
* Histopathologic diagnosis of glioma or glioneuronal tumor.
* At least one measurable lesion as defined by RANO criteria.
* Meet indication for first-line systemic therapy.

Exclusion Criteria:

* Participant has any of the following tumor-histological findings:

  1. Schwannoma
  2. Subependymal giant cell astrocytoma (Tuberous Sclerosis)
  3. Diffuse intrinsic pontine glioma, even if histologically diagnosed as World Health Organization (WHO) Grade I-II
* Participant's tumor has additional pathogenic molecular alterations, including but not limited to a) isocitrate dehydrogenase (IDH) 1/2 mutation, b) Histone H3 mutation, and c) neurofibromatosis Type 1 (NF-1) loss of function alteration.
* Known or suspected diagnosis of NF-1/ neurofibromatosis Type 2 (NF-2).
* Prior or ongoing nonsurgical anticancer therapy for this indication (eg, chemotherapy, oral/IV targeted therapy) including radiation.

Max Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 400 (Estimated)
Dates: Start 2023-02-27 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2030-03 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) of tovorafenib monotherapy versus SoC chemotherapy | Up to 60 months
  ORR assessed per Response Assessment in Pediatric Neuro Oncology (RAPNO) criteria by Independent Review Committee (IRC), and defined as the proportion of participants with overall confirmed response of complete response (CR), partial response (PR), or minor response (MR).

SECONDARY OUTCOMES:
Progression-free survival (PFS) of tovorafenib monotherapy versus SoC chemotherapy | Up to 60 months
  PFS assessed per RAPNO criteria by IRC, and deﬁned as time from randomization to PD or death from any cause, whichever comes first.
Event-free survival (EFS) of tovorafenib monotherapy versus SoC chemotherapy | Up to 60 months
  EFS assessed per RAPNO criteria by IRC, deﬁned as time from randomization to PD, death from any cause, or initiation of any new anticancer therapy, whichever comes first.
Overall survival (OS) of tovorafenib monotherapy versus SoC chemotherapy | Up to 60 months
  Overall survival is defined as time from randomization up to death from any cause.
Number of participants with any treatment-emergent adverse events, and Serious adverse events | Up to 60 months
  Type, frequency, and severity of adverse events of tovorafenib monotherapy versus SoC chemotherapy will be assessed.
. Number of participants with clinically significant vital signs and laboratory abnormalities findings | Up to 60 months
  Type, frequency, and severity of vital signs and laboratory abnormalities of tovorafenib monotherapy versus SoC chemotherapy will be assessed.
Change from baseline in Adaptive Behavior Composite Score (ABS) of tovorafenib monotherapy versus SoC chemotherapy | Baseline, Year 1, 2 and 5
  Adaptive behavior Composite Score will be evaluated using domain scores collected from the comprehensive Vineland III Adaptive Behavior Scale (VABS).
Change from baseline in the Motor Skills Domain Score of tovorafenib monotherapy versus SoC chemotherapy | Baseline, Year 1, 2 and 5
  The motor skills (gross and fine) will be assessed using the Motor Skills Score domain of the VABS in pediatric participants.
Change from baseline in the Daily Living Domain Score of tovorafenib monotherapy versus SoC chemotherapy | Baseline, Year 1, 2 and 5
  The daily living (personal, domestic and community) will be assessed using Daily Living Domain Score of VABS.
Change from baseline in the Communication Domain Score of tovorafenib monotherapy versus SoC chemotherapy | Baseline, Year 1, 2 and 5
  The communication skills (receptive, expressive and written) will be assessed using Communication Domain Score of VABS.
Change from baseline in the Socialization Domain Score of tovorafenib monotherapy versus SoC chemotherapy | Baseline, Year 1, 2 and 5
  The socialization skills (Interpersonal relationships, play and leisure time and coping skills) will be assessed using Socialization Domain Score of VABS.
Change in age-adjusted visual acuity (VA) of tovorafenib monotherapy versus SoC chemotherapy in optic pathway glioma (OPG) participants aged < 3 years | Baseline and up to 5 years
  Visual acuity testing using current age-appropriate testing methodology will be performed for all participants at Screening. For participants with OPG or an underlying visual deficit related to the primary malignancy, visual acuity testing will be performed every time participants have a radiographic response assessment. Assessments will be performed in each eye separately at a recommended testing distance of 3 meters.
Change in best corrected visual acuity of tovorafenib monotherapy versus SoC chemotherapy in OPG participants aged ≥ 3 years | Baseline and up to 5 years
  Visual acuity assessments to be performed by an ophthalmologist or another qualified site clinical personnel.
Visual progression-free survival (v-PFS) of tovorafenib monotherapy versus SoC chemotherapy | Up to 60 months
  Visual progression-free survival is defined as the time from start of treatment to visual event for OPG participants aged ≥ 3 years.
ORR of tovorafenib monotherapy versus SoC chemotherapy | Up to 60 months
  ORR, defined as the proportion of participants with overall confirmed response per Response Assessment in Neuro-Oncology for High-Grade Glioma (RANO-HGG) criteria (CR or PR) and RANO-LGG criteria (CR, PR, or MR), as applicable.
Clinical beneﬁt rate (CBR) of tovorafenib monotherapy versus SoC chemotherapy | Up to 60 months
  CBR, deﬁned as the proportion of participants with radiological tumor stabilization or regression per RANO-LGG (CR, PR, MR, or SD lasting 12 months or more), RANO-HGG (CR, PR, or SD lasting 12 months or more) or RAPNO criteria (CR, PR, MR or SD lasting 12 months or more), as applicable.
Time to response (TTR) of tovorafenib monotherapy versus SoC chemotherapy | Up to 60 months
  TTR, measured by the time following randomization to ﬁrst imaging of tumor response that was subsequently conﬁrmed per RANO-HGG criteria (CR or PR), RANO-LGG criteria (CR, or PR, or MR), or RAPNO criteria (CR, PR, or MR), as applicable.
PFS of tovorafenib monotherapy versus SoC chemotherapy | Up to 60 months
  PFS per RANO-HGG or RANO-LGG criteria (as applicable), deﬁned as time from randomization to PD or death from any cause, whichever occurs first.
EFS of tovorafenib monotherapy versus SoC chemotherapy | Up to 60 months
  EFS per RANO-HGG or RANO-LGG criteria (as applicable), defined as time from randomization to PD, death from any cause, or initiation of any new anticancer therapy, whichever comes first.
Duration of response (DOR) of tovorafenib monotherapy versus SoC chemotherapy | Up to 60 months
  DOR, deﬁned as time from first imaging of tumor response per RANO-LGG, RANO-HGG or RAPNO criteria, as applicable, that was subsequently confirmed to radiographic PD or death from any cause, whichever comes first.
Change from Baseline in health-related quality of life (HRQoL) total score of tovorafenib monotherapy versus SoC chemotherapy | Baseline, Year 1, 2 and 5
  The Patient-Reported Outcomes Measurement Information System (PROMIS®) Pediatric/Parent Proxy Profile 49 v2.0 will be used to assess mental and social HRQoL.

CONTACTS AND LOCATIONS:
Locations (138):
- United States (38):
  - Children's of Alabama, Birmingham, Alabama
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Children's Hospital Los Angeles, Los Angeles, California
  - Children's Hospital of Orange County Main Campus - Orange, Orange, California
  - Packard Children's Hospital Stanford, Palo Alto, California
  - UCSF Benioff Children's Hospital, San Francisco, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Children's National Medical Center, Washington D.C., District of Columbia
  - University of Florida Health, Gainesville, Florida
  - Nicklaus Children's Hospital, Miami, Florida
  - Arnold Palmer Hospital for Children, Orlando, Florida
  - Johns Hopkins All Children's Hospital, St. Petersburg, Florida
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Riley Hospital for Children at Indiana University Health, Indianapolis, Indiana
  - University of Iowa Hospitals Clinics, Iowa City, Iowa
  - Norton Children's Hospital, Louisville, Kentucky
  - Maine Children's Cancer Program, Scarborough, Maine
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan - - C.S. Mott Children's Hospital, Ann Arbor, Michigan
  - Children's Minnesota, Minneapolis, Minnesota
  - Childrens MS Cncr Ctr Bld Dsr, Jackson, Mississippi
  - St. Louis Children's Hospital, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Albany Medical Center, Albany, New York
  - New York University Langone Health, New York, New York
  - Columbia University, New York, New York
  - University of Rochester, Rochester, New York
  - Duke Cancer Institute, Durham, North Carolina
  - Cleveland Clinic Main Campus, Cleveland, Ohio
  - Oregon Health Science University, Portland, Oregon
  - Dell Children's Medical Center of Central Texas, Austin, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Texas Children's Hospital, Houston, Texas
  - Seattle Children's Hospital, Seattle, Washington
  - University of Wisconsin - Madison, Madison, Wisconsin
- Australia (6):
  - Children's Health Queensland Hospital and Health Service, South Brisbane, Queensland
  - Perth Children's Hospital, Nedlands
  - Women's and Children's Health Network, North Adelaide
  - The Royal Children's Hospital - Children's Cancer Centre, Parkville
  - Sydney Children's Hospital - Randwick, Randwick
  - Children's Hospital at Westmead, Westmead
- Austria (2):
  - Medizinische Universität Innsbruck, Innsbruck, Tyrol
  - Medizinische Universität Wien, Vienna
- Belgium (3):
  - Cliniques Universitaires Saint-Luc, Brussels
  - Universitair Ziekenhuis Gent, Ghent
  - Universitair Ziekenhuis Leuven - Campus Gasthuisberg, Leuven
- Grupo de Apoio ao Adolescente e à Criança com Câncer (GRAACC), São Paulo, Brazil
- Canada (10):
  - Alberta Children's Hospital, Calgary, Alberta
  - Stollery Children's Hospital, Edmonton, Alberta
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - McMaster Children's Hospital, Hamilton, Ontario
  - Children's Hospital London Health Sciences Centre, London, Ontario
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - CHU Sainte-Justine, Montreal, Quebec
  - The Montreal Children's Hospital, Montreal, Quebec
  - Centre Hospitalier de l'Université Laval et Centre Mère-Enfant Soleil, Québec
  - SickKids - The Hospital for Sick Children, Toronto
- Czechia (2):
  - Fakultní Nemocnice Brno - D?tská Nemocnice, Brno
  - Motol University Hospital, Prague
- Denmark (2):
  - Aarhus Universitetshospital, Aarhus, Central Jutland
  - Rigshospitalet, Copenhagen
- CCHE, Cairo, Cairo Governorate, Egypt
- Finland (2):
  - Helsingin yliopistollinen sairaala (HUS), Helsinki
  - Tampereen Yliopistollinen Sairaala, Tampere
- France (5):
  - Centre de Lutte contre le Cancer - Centre Oscar Lambret, Lille
  - Centre Léon Bérard, Lyon
  - Hôpital de la Timone, Marseille
  - Institut Curie, Paris
  - Gustave Roussy, Villejuif
- Germany (13):
  - Universitätsklinikum Freiburg, Freiburg im Breisgau, Baden-Wurttemberg
  - Universitätsklinikum Augsburg, Augsburg, Bavaria
  - Universitätsklinikum Erlangen, Erlangen, Bavaria
  - Universitätsklinikum Würzburg, Würzburg, Bavaria
  - Universitätsklinikum Frankfurt, Frankfurt am Main, Hesse
  - Medizinische Hochschule Hannover, Hanover, Lower Saxony
  - Universitaetsklinikum Essen, Essen, North Rhine-Westphalia
  - Universitätsklinikum Leipzig, Leipzig, Saxony
  - Charité Universitätsmedizin Berlin, Berlin
  - Evangelische Klinikum Bethel (EvKB), Bielefeld
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg
  - Universitätsklinikum Heidelberg, Heidelberg
  - Universitätsklinikum Tübingen, Tübingen
- Greece (2):
  - Aghia Sofia General Children's Hospital, Athens
  - Athens General Children's Hospital, Athens
- Semmelweis Egyetem Tűzoltó utcai II. Sz. Gyermekgyógyászati Kliniká, Budapest, Hungary
- Children's Health Ireland at Crumlin, Crumlin, Dublin, Ireland
- Israel (2):
  - Schneider Children's Medical Center of Israel, Petah Tikva
  - The Edmond and Lily Safra Children's Hospital, Ramat Gan
- Italy (9):
  - Fondazione IRCCS - Istituto Nazionale dei Tumori, Milan, Milan
  - Ospedale Pediatrico Bambino Gesù, Roma, Rome
  - Ospedale Infantile Regina Margherita, Torino, Turin
  - Azienda Universitaria Ospedaliera Consorziale - Policlinico di Bari, Bari
  - Azienda Ospedaliera U. Meyer, Florence
  - Istituto Giannina Gaslini, Genova
  - Azienda Ospedaliera di Rilievo Nazional Santobono Pausilipon, Napoli
  - Azienda Ospedale Università di Padova, Padua
  - Azienda Sanitaria Universitaria Friuli Centrale - P.O. Santa Maria della Misericordia, Udine
- King Hussein Cancer Foundation - King Hussein Cancer Center, Amman, Muhafazat al-Asima, Jordan
- Prinses Maxima Centrum Kinderoncologie, Utrecht, Netherlands
- Starship Paediatric Blood & Cancer Center, Grafton, New Zealand
- Norway (2):
  - Universitetssykehuset Nord-Norge - Tromsø, Tromsø, Troms
  - Oslo Universitetssykehus, Oslo
- Sidra Medicine, Doha, Qatar
- SingHealth Group - KK Women's and Children's Hospital, Singapore, Singapore
- Univerzitetni Klinini Center Ljubljana, Ljubljana, Slovenia
- South Korea (2):
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Seoul
- Spain (7):
  - Hospital Universitario Cruces, Barakaldo
  - Hospital Universitari Vall d'Hebrón, Barcelona
  - Hospital Sant Joan de Déu Barcelona, Barcelona
  - Hospital Infantil Universitario Niño Jesús, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Virgen del Rocío, Seville
  - Hospital Universitari i Politècnic La Fe, Valencia
- Sweden (3):
  - Drottning Silvias barn- och ungdomssjukhus, Gothenburg
  - Skånes Universitetssjukhus - Lund, Lund
  - Astrid Lindgrens Barnsjukhus Solna, Stockholm
- Switzerland (2):
  - Centre Hospitalier Universitaire Vaudois Lausanne, Lausanne
  - Universitaets - Kinderspital Zürich, Zurich
- Taiwan (2):
  - Taipei Medical University Hospital, Taipei
  - Chang Gung Memorial Hospital - Linkou Branch, Taoyuan District
- United Kingdom (14):
  - Birmingham Women's and Children's NHS Foundation Trust, Birmingham, England
  - Leeds Teaching Hospital NHS Trust, Leeds, England
  - Alder Hey Children's NHS Foundation Trust, Liverpool, England
  - Manchester University NHS Foundation Trust, Manchester, England
  - The Newcastle Upon Tyne Hospitals NHS Foundation Trust, Newcastle upon Tyne, England
  - Great Ormond Street Hospital for Children, Oxford, England
  - University Hospital Southampton NHS Foundation Trust, Southampton, Hampshire
  - Royal Belfast Hospital for Sick Children, Belfast, Northern Ireland
  - NHS Greater Glasgow and Clyde, Glasgow, Scotland
  - Sheffield Children's Hospital, Sheffield, South Yorkshire
  - The Royal Marsden NHS Foundation Trust, Sutton, Surrey
  - University Hospitals Bristol and Weston NHS Foundation Trust, Bristol
  - Cambridge University Hospitals NHS Foundation Trust, Cambridge
  - The Christie Hospital, Manchester

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] van Tilburg CM, Kilburn LB, Perreault S, Schmidt R, Azizi AA, Cruz-Martinez O, Zapotocky M, Scheinemann K, Meeteren AYNS, Sehested A, Opocher E, Driever PH, Avula S, Ziegler DS, Capper D, Koch A, Sahm F, Qiu J, Tsao LP, Blackman SC, Manley P, Milde T, Witt R, Jones DTW, Hargrave D, Witt O. LOGGIC/FIREFLY-2: a phase 3, randomized trial of tovorafenib vs. chemotherapy in pediatric and young adult patients with newly diagnosed low-grade glioma harboring an activating RAF alteration. BMC Cancer. 2024 Jan 30;24(1):147. doi: 10.1186/s12885-024-11820-x. PMID 38291372